CLINICAL TRIAL: NCT06425705
Title: Evaluating the Outcome of Silymarin as an Adjunct Therapy to Renin-Angiotensin System Inhibitors in Proteinuric Type 2 Diabetic Patients
Brief Title: Impact of Silymarin Adjunct Therapy on Proteinuria in Type 2 Diabetic Patients on RAS Inhibitors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lahore General Hospital (Other Government)
Responsible Party: Principal Investigator, Muhammad Irfan Jamil, Principal Investigator, Lahore General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LahoreGeneralH1
Record Dates: First submitted 2024-05-07; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Proteinuria; Type 2 Diabetes Mellitus; Renin-Angiotensin System
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Proteinuria | interventions — Silymarin; milk-thistle extract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Silymarin (Experimental): Received 140 mg of silymarin administered orally three times daily, alongside their standard treatment with renin-angiotensin system inhibitors.
  Interventions: Drug: Silymarin
- Group Placebo (Placebo Comparator): Received placebo capsule three times a day alongside their standard treatment with renin-angiotensin system inhibitors.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Silymarin — 140 mg of silymarin administered orally three times daily, alongside their standard treatment with renin-angiotensin system inhibitors.
  Other Names: Milk thistle extract
  Arms: Group Silymarin
Drug: Placebo — placebo capsule three times a day alongside their standard treatment with renin-angiotensin system inhibitors.
  Arms: Group Placebo

SUMMARY:
Given the inadequacies of existing pharmacological interventions for diabetic nephropathy, this study is predicated on the hypothesis that silymarin, having shown promise in mitigating hyperglycemia in diabetic patients without nephropathy and displaying renal protective effects in animal models, merits a thorough and systematic investigation. The current body of research on silymarin, particularly human trials, is limited by small cohorts and the preliminary nature of its outcomes. This research aims to evaluate the efficacy of silymarin as an adjunctive treatment in patients with Type 2 diabetes mellitus (T2DM) already on renin-angiotensin system inhibitors, focusing on its potential to reduce proteinuria and improve renal function. The ultimate objective is to amass more definitive evidence that could potentially inform a new therapeutic approach in the management of diabetic nephropathy.

DETAILED DESCRIPTION:
After securing the approval from the Ethical Review Board of hospital, this study was conducted in the Nephrology Department, Lahore General Hospital, Lahore. All patients diagnosed with Type 2 Diabetes Mellitus was assessed based on the previously defined inclusion and exclusion criteria. Informed consent was obtained from all eligible participants who agreed to participate in the study.

Baseline Data Collection: Upon enrollment, demographic and clinical information including age, gender, duration of diabetes, baseline renal function tests, current medication use, and baseline measures of HBA1c, FBS, RBS and proteinuria were collected. This information was provided a comprehensive profile of each participant at the start of the study.

Treatment Allocation: Patients was randomly assigned into two groups using a lottery method:

* Group A: received 140 mg of silymarin administered orally three times daily, alongside their standard treatment with renin-angiotensin system inhibitors.
* Group B: received placebo capsule three times a day alongside their standard treatment with renin-angiotensin system inhibitors.

Monitoring and Follow-up Assessments: Participants was assessed for outcomes after at one month and 3 months to monitor changes in proteinuria and renal function. Specific tests were included:

* Measurement of Urinary Albumin-Creatinine Ratio (UACR): Participants were required to provide 24-hour urine specimens at one month and three months into the study. To ensure that the urine samples are not affected by external factors, patients was instructed to maintain their usual physical activities and avoid strenuous exercises the evening before the assessment days. Proteinuria was quantified using immunoturbidimetry.
* Assessment of Serum Creatinine and Calculation of eGFR to Monitor Renal Function: The estimated glomerular filtration rate (eGFR) was calculated using the CKD-EPI formula at one month and three months. These assessments were help to monitor any changes in renal function over the course of the study.
* Measurement of HbA1c levels after 3 months. The data was recorded meticulously using standardized data collection forms. Data was analyzed using SPSS version 26.0. Baseline characteristics of participants (age, gender, duration of diabetes, baseline renal function tests, HbA1c, FBS, RBS) were summarized using means and standard deviations for continuous variables, and frequencies and percentages for categorical variables. Changes in UACR, eGFR, and HbA1c from baseline to one month and three months were compared between Group A (silymarin) and Group B (placebo) using independent t-tests or Mann-Whitney U tests, depending on the normality of the data. Analysis of Covariance (ANCOVA) was used to adjust for any baseline imbalances and potential confounders between the two groups. Repeated measures ANOVA were employed to analyze changes over time within and between treatment groups for UACR, eGFR, and HbA1c levels, accounting for within-subject correlation over the assessment periods. All statistical tests were two-sided, and a p-value of less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 35-70 years.
* Both male and female with Type II diabetes.
* Overt proteinuria defined by urinary albumin excretion > 300 mg/24 hr. in 2 consecutive determinations despite treatment with highest FDA recommended doses of an angiotensin converting enzyme inhibitor or angiotensin receptor blocker for at least 6 months.
* Treatment of hyperglycemia with (but not limited to) an oral hypoglycemic agent or insulin (If a SGLT2 inhibitors is used, stable dose for at least 3 months).
* Treatment of hypercholesterolemia with (but not limited to) one medication from the class statins.
* Patients using stable dose of Non-Dihydropyridine Calcium Channel Blockers for at least 6 months as antihypertensive.
* Presence of diabetic retinopathy.
* Signing informed consent.

Exclusion Criteria:

* Type I diabetes.
* Advanced chronic kidney disease defined by estimated GFR < 30 ml/min/1.73 m2
* Severely uncontrolled diabetes defined by HbA1C > 10%.
* Uncontrolled hypertension defined by SBP >140 mmHg or DBP >90 mmHg despite antihypertensive therapy.
* Patients with organ transplant history.
* Secondary forms of hypertension with defined etiology other than diabetes mellitus.
* Other renal diseases.
* Chronic Heart Failure with NYHA class III or IV.
* Active infection.
* Pregnancy.

Use of one of the following medications within 2 months prior to enrollment in the study:

* Non-steroidal anti-inflammatory agents.
* Antioxidants supplements including vitamin E, vitamin C, N-acetyl- cysteine (NAC), Pentoxifylline, Lipoic acid, Fish-oil extracts (omega-3 fatty acids), Soy extracts (isoflavones), Green-tea preparations, Pomegranate extracts, Grape extracts.
* Active malignancy.
* History of drug or alcohol dependency.
* Psychiatric or neurological condition, preventing aware consent to the study and/or adherence to the study protocol.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Change in the urinary albumin-creatinine ratio (UACR) from baseline | Outcomes monitored at one and three-month intervals
  It was measured quantitatively by comparing the urinary albumin-creatinine ratio (UACR) in mg/g between initial recruitment and subsequent follow-up visits at one and three months.
Change in estimated glomerular filtration rate (eGFR) from baseline | Outcomes monitored at one and three-month intervals
  eGFR was calculated using the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) formula, which incorporates serum creatinine, age, sex, and race. The outcome measure was the change in eGFR in mL/min/1.73 m² at one month and three months compared to the baseline value.
Change in HbA1c levels from baseline | Outcomes monitored after three-month.
  It was measured quantitatively by comparing the HbA1c levels in percentage (%) between initial recruitment and subsequent follow-up visit after three months.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Irfan Jamil, MBBS, FCPS, Principal Investigator — Lahore General Hospital, Lahore
Locations (1):
- Lahore General Hospital, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
will be shared on special request